CLINICAL TRIAL: NCT00432835
Title: Double-Blind Placebo-Controlled Cross-Over Design With Wash-Out for Temporary Gastric Electrical Stimulation for Drug Refractory Gastroparesis
Brief Title: Temporary Gastric Electrical Stimulation for Drug Refractory Gastroparesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Thomas Abell, MD, Principal Investigator, Professor of Medicine, Director, Division of Digestive Diseases, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-0185
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Gastroparesis
Keywords: Nausea; Vomiting; Delayed gastric emptying; Diabetes Mellitus; Post-Surgical; Idiopathic
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastric Stimulation Days1-4/Sham5-8 (Active Comparator): The sequence followed for patients in Group 1 was: enrollment and acquisition of baseline data, then placement of electrode, then determination of mucosal EGG, then randomization to Group 1, then active stimulation for 72 consecutive hours, then a 1 day wash out, then the cross over, which entailed the device remaining inactive for the final 3 study days
  Interventions: Device: Gastric Electrical Stimulator, Enterra, Medtronics, Inc.
- Sham1-4/Gastric Stimulation Days5-8 (Active Comparator): The sequence followed for patients in Group 2 was: enrollment and acquisition of baseline data, then placement of electrode, then determination of mucosal EGG, then randomization to Group 2, then no stimulation whatsoever until Day 5, then the cross over,then active stimulation with the Gastric Electrical Stimulator for 72 consecutive hours.
  Interventions: Device: Gastric Electrical Stimulator, Enterra, Medtronics, Inc.

INTERVENTIONS:
Device: Gastric Electrical Stimulator, Enterra, Medtronics, Inc. — All patients received a GES electrode, endoscopically placed and connected to an external device at baseline. The device was turned ON to provide 72 continuous hours of active stimulation and OFF to deactivate stimulation
  Other Names: No other name currently exists.

SUMMARY:
The purpose of this research is to determine if temporary gastric electrical stimulation will help improve symptoms of gastroparesis (abnormal stomach emptying). We hypothesize that when the device is ON, Gastrointestinal symptoms will decrease by at least 50% from baseline.

DETAILED DESCRIPTION:
Gastric Electrical Stimulation is an established treatment for drug-refractory patients who have the symptoms of gastroparesis/gastropathy. The symptoms of GP are nausea, vomiting, anorexia/early satiety, bloating/distention and abdominal pain and are classically associated with delayed gastric emptying of solids. The technique of GES was first used, in a patient seen at University of Tennesse-Memphis in 1993 and has undergone several clinical trials, particularly the GEMS trial, a feasibility trial starting in 1995 and the WAVESS trial, a double-blind trial begun in 1997. Both were international trials, showing promising results, and both have been published in the last 2 years. However, a number of issues related to who would benefit the most from Gastric Electrical Stimulation therapy have emerged. Among these issues are whether patients with etiologies other than diabetic or idiopathic gastroparesis, such as post-surgical gastropathy, which is often related to rapid, not delayed gastric emptying could be helped.

Most recently a technique for the temporary placement of a Gastric Electrical Stimulation electrode in the stomach with an upper endoscope, combined with an external Gastric Electrical Stimulation device, has been tried and validated, first at UAMS in Little Rock, AR, beginning in 2001 and more recently here at UMMC, beginning later in 2001 and up until the present time. Using the technique of temporary gastric electrical stimulation, we have been able to demonstrate that TempStim can quickly demonstrate (in a manner of days) that a patient will respond to temporary GES, as quantified by a decrease in GI total symptoms and an improvement and normalization in solid gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male of Female
* Age Range: 18 to 70 inclusive
* Patients with GP of diabetic, surgically related or idiopathic etiology.
* Symptoms of GP for >/= 1 year.
* Refractory or intolerant to antiemetic drug classes (antihistamines and phenothiazines, serotonin receptor antagonists, dopamine receptor antagonists)
* Chronic vomiting and/or nausea with 7 or more episodes per week for either symptom irrespective of GET values.
* The patient is willing and able to provide informed consent.
* The patient is willing and able to return for required follow-up visits.

Exclusion Criteria:

* Patients < 18 or >70 years in age.
* Patients with an active infection of any kind.
* Patients who the investigator determines are not candidates for endoscopic procedures.
* Women who are pregnant
* Inability or unwillingness to provide informed consent
* Unwilling or unable to return for required follow-up visits and examinations.
* Patients who are currently enrolled in another investigation of a medical device or drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Abell, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Result] Abell TL, Johnson WD, Kedar A, Runnels JM, Thompson J, Weeks ES, Minocha A, Griswold ME. A double-masked, randomized, placebo-controlled trial of temporary endoscopic mucosal gastric electrical stimulation for gastroparesis. Gastrointest Endosc. 2011 Sep;74(3):496-503.e3. doi: 10.1016/j.gie.2011.05.022. PMID 21872708
- See also: Pub Med abstract of study as reported in "Gastrointestinal Endoscopy" — http://www.ncbi.nlm.nih.gov/pubmed?term=%22Gastrointestinal+endoscopy%22%5BJour%5D+AND+74%5Bvolume%5D+AND+3%5Bissue%5D+AND+496%5Bpage%5D+AND+2011%5Bpdat%5D+AND+Abell%5Bfirst+author%5D+AND+double-masked&TransSchema=title&cmd=detailssearch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seeking temporary gastric electric stimulator devices for drug-refractory gastroparesis between August 2005 and October 2006 who met the inclusion criteria and did not have any of the exclusion criteria were offered access to the research protocol.
Pre-assignment Details: No significant events or approaches for the overall study following participant enrollment were performed prior to group assignment.
Groups:
- Gastric Stimactivated Days1-4/Not Activated Days5-8: The sequence followed for patients in Group 1 was: enrollment and acquisition of baseline data, then placement of electrode, then determination of mucosal Electrogastrogram, then randomization to Group 1, then active stimulation for 72 consecutive hours, then a 1 day wash out, then the cross over, which entailed the device remaining inactive for the final 3 study days
- Gastric StimulationNotActivated Days1-4/Activated Days5-8: The sequence followed for patients in Group 2 was: enrollment and acquisition of baseline data, then placement of electrode, then determination of mucosal EGG, then randomization to Group 2, then no stimulation whatsoever until Day 5, then the cross over,then active stimulation with the Gastric Electrical Stimulator for 72 consecutive hours.
Period: Overall Study
Arm/Group | Gastric Stimactivated Days1-4/Not Activated Days5-8 | Gastric StimulationNotActivated Days1-4/Activated Days5-8
Started | 28 | 30
Completed 1st Intervention | 22 | 23
Completed 2nd Intervention | 22 | 23
Completed | 22 (These 22 patients completed the entire 8 day protocol.) | 23 (These 23 patients completed the entire 8 day protocol.)
Not Completed | 6 | 7
Not completed — Adverse event: lead dislodgement. | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Stimactivated Days1-4/Not Activated Days5-8 | Gastric StimulationNotActivated Days1-4/Activated Days5-8 | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 2 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 47 (14) | 47 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Symptom of Vomiting Associated With Gastroparesis
Description: Likert Scale 0-4 (low-high) using a patient reported outcomes tool
Time Frame: Study Day 0 (Baseline), Day 3, Day 7
Measure: Mean (Standard Error); unit: Patient Self-reported Symptom Score
Groups:
- Gastric StimulationNotActivated Days1-4/Activated Days5-8: The sequence followed for patients in Group 2 was: enrollment and acquisition of baseline data, then placement of electrode, then determination of mucosal electrogastrogram, then randomization to Group 2, then no stimulation whatsoever until Day 5, then the cross over,then active stimulation with the Gastric Electrical Stimulator for 72 consecutive hours.
Arm/Group | Gastric Stimactivated Days1-4/Not Activated Days5-8 | Gastric StimulationNotActivated Days1-4/Activated Days5-8
Number analyzed (Participants) | 28 | 30
Patient Self-reported Symptom Score
  Vomiting Score Day 0 | 1.82 (1.55) | 2.68 (1.61)
  Vomiting Score Day 3 | 0.17 (0.67) | 1.20 (1.47)
  Vomiting Score Day 7 | 0.91 (1.44) | 0.72 (1.17)

2. Primary Outcome: Symptom of Nausea Associated With Gastroparesis
Description: Likert Scale 0-4 (low-high) using a patient reported outcomes tool
Time Frame: Study Day 0 (Baseline), Day 3, Day 7
Measure: Mean (Standard Error); unit: Patient Self-reported Symptom Score
Arm/Group | Gastric Stimactivated Days1-4/Not Activated Days5-8 | Gastric StimulationNotActivated Days1-4/Activated Days5-8
Number analyzed (Participants) | 28 | 30
Patient Self-reported Symptom Score
  Nause Score Day 0 | 3.27 (0.92) | 3.33 (1.03)
  Nausea Score Day 3 | 1.46 (1.29) | 1.67 (1.49)
  Nausea Score Day 7 | 2.26 (1.18) | 1.4 (1.38)

3. Primary Outcome: Symptom of Gastric Emptying Time (GET) Associated With Gastroparesis
Description: Transit time of a radio-labeled meal through the stomach, measured by scintigraphy for %contents remaining in the stomach at 1 hour, 2 hours, and 4 hours. GET measures were obtained at baseline, during the period allowed for 'washout', and on the final study day.
Time Frame: Study Day 0 (Baseline), Day 4, Day 8
Measure: Mean (Standard Error); unit: percentage of radiolabeled meal in stoma
Arm/Group | Gastric Stimactivated Days1-4/Not Activated Days5-8 | Gastric StimulationNotActivated Days1-4/Activated Days5-8
Number analyzed (Participants) | 28 | 30
percentage of radiolabeled meal in stoma
  GET Day 0, at 1st hour | 67.07 (20.23) | 66.13 (25.37)
  GET Day 0, at 2nd hour | 69.96 (23.79) | 37.41 (28.06)
  GET Day 0, at 4th hour | 64.71 (21.10) | 16.43 (23.00)
  GET Day 4, at 1st hour | 69.96 (23.79) | 62.35 (24.75)
  GET Day 4, at 2nd hour | 46.85 (25.30) | 38.00 (24.64)
  GET Day 4, at 4th hour | 24.11 (23.76) | 21.85 (28.51)
  GET Day 8, at 1st hour | 64.71 (21.10) | 68.67 (19.92)
  GET Day 8, at 2nd hour | 42.19 (24.37) | 40.92 (26.50)
  GET Day 8, at 4th hour | 24.71 (27.94) | 20.25 (25.26)

ADVERSE EVENTS:
Time Frame: Study Days 0-8 (Entirety of Study)
Groups:
- Gastric Stimactivated: Gastric Electrical Stimulation
- Gastric StimulationNotActivated: Sham stimulation
Arm/Group | Gastric Stimactivated | Gastric StimulationNotActivated
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 6/51 | 7/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Stimactivated (N=51) | Gastric StimulationNotActivated (N=52)
Lead Dislodgment (Gastrointestinal disorders) | 6 (6) | 7 (7) — All lead dislodgment occurred by Day 4.

LIMITATIONS AND CAVEATS:
New lead implantation techniques now minimize dislodgment (only adverse effect); Parallel, non-crossover protocol will address any carry-over effect after tGES activation OFF; stratification for baseline mucosal EGG and medications may be useful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes